CLINICAL TRIAL: NCT02721875
Title: An Open Label, Phase I Trial of Intravenous Administration of Volasertib as Monotherapy and in Combination With Azacitidine in Patients With Myelodysplastic Syndrome After Hypomethylating Agents Treatment Failure
Brief Title: Trial of Volasertib With or Without Azacitidine in Patients With Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1230.43; 2015-004490-32 (EudraCT Number)
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Results first posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — BI 6727; Azacitidine

ARMS (2):
- Volasertib monotherapy (Experimental)
  Interventions: Drug: Volasertib
- Volasertib + azacitidine combination (Experimental)
  Interventions: Drug: Volasertib; Drug: Azacitidine

INTERVENTIONS:
Drug: Volasertib
  Arms: Volasertib monotherapy
Drug: Volasertib
  Arms: Volasertib + azacitidine combination
Drug: Azacitidine
  Arms: Volasertib + azacitidine combination

SUMMARY:
The objectives of this trial are to evaluate the safety, tolerability, maximum tolerated dose (MTD), pharmacokinetics and preliminary efficacy of volasertib in two dosing schedules of intravenous volasertib as monotherapy or in combination with azacitidine in patients with myelodysplastic syndrome (MDS) after hypomethylating agents (HMA) treatment failure.

ELIGIBILITY:
Inclusion criteria:

* Patients 18 years and older with diagnosis of WHO classification-defined primary or treatment-related myeloid neoplasms classified as follows:
* Refractory anaemia with excess blasts (RAEB)-1 (5%-9% marrow blasts) or
* RAEB-2 (10%-19% marrow blasts or 5% - 19% peripheral blast) or
* Chronic Myelomonocytic Leukaemia (CMML) (5%-19% blasts) with white blood cell (WBC) count <13000/mm3 or
* Acute Myeloid Leukaemia (AML) (20%-29% marrow blasts, i.e., RAEB-t according to French-American-British [FAB] classification) with WBC count <10000/mm3
* Patients classified as intermediate, high or very high-risk according to Revised - International Prognostic Scoring System (IPSS-R) at the time of enrolment
* Patients who have received a maximum of 24 cycles of frontline HMA treatment prior to enrolment.
* Patients must have received a minimum prior dosing schedule of either:
* Azacitidine 75 mg/m2 x 5 days per cycle or 50 mg/m2 x 7 days per cycle, or
* Decitabine 20 mg/m2 x 5 days per cycle, or
* SGI-110 60 mg/m2 x 5 days per cycle
* Patients must meet either one of the following criteria:
* Progressive disease (PD, according to 2006 International Working Group (IWG) criteria) at any time after initiation of the prior HMA treatment, or
* Relapse after initial complete (CR) or partial remission (PR) or haematological improvement (HI) (according to 2006 IWG criteria); or
* Failure to achieve complete or partial remission or HI (according to 2006 IWG) with no evidence of progression (i.e., Stable Disease [SD]) after at least six cycles of prior azacitidine treatment or at least four cycles of other prior HMA treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2 at screening
* Signed written informed consent consistent with International Conference of Harmonization Good Clinical Practice (ICH-GCP) and local legislation

Exclusion criteria:

* Prior systemic therapy (including investigational drugs) for MDS, CMML or AML within 14 days before treatment with study medication.
* Patients requiring intervention for white blood cell count control with hydroxyurea, chemotherapy, or leukapheresis.
* Prior exposure to more than one line of HMA based treatment.
* Prior exposure to volasertib or other polo-kinase inhibitors
* Patients who were unable to tolerate prior HMA treatment
* Patients with history of hematopoietic stem cell transplant (HSCT)
* Known hypersensitivity to the trial drugs or its excipients
* Second malignancy currently requiring active therapy (except for hormonal/anti-hormonal treatment, e.g., in prostate or breast cancer).
* QTcF value >470 ms or QT prolongation deemed clinically relevant by the investigator (e.g., congenital long QT syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2016-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- University of Fukui Hospital, Fukui, Yoshida-gun, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Volasertib Monotherapy: Subject received volasertib with starting dose of 110 mg/meter square (m2) in solution for intravenous infusion (350 milligram (mg)/175 milliliter (mL) vial (2.0 mg/mL)), on day 1 + 8, 28-day cycle
- Volasertib + Azacitidine Combination: Subject received volasertib with starting dose 170 mg/m2 on day 8 in combination with subcutaneous (s.c.) or intravenous administration of azacitidine 75 mg/m2 once daily for 7 consecutive days (days 1-7), 28-day cycle
Period: Overall Study
Arm/Group | Volasertib Monotherapy | Volasertib + Azacitidine Combination
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Progressive disease/relapse | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients who were documented to receive at least one dose of volasertib were defined as the treated set (TS).
Groups:
- Total: Total of all reporting groups
Arm/Group | Volasertib Monotherapy | Volasertib + Azacitidine Combination | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69 |  | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities (DLT) in the First Cycle
Description: DLT was defined as any of the following adverse events (AEs) considered to be related to study drug: 1. Common terminology criteria for adverse events (CTCAE) v4.03 ≥Grade 3 drug related non- haematological toxicity, excluding; ≥Grade 3 untreated nausea, vomiting or diarrhea. Any laboratory abnormality - not considered clinically significant by investigator or resolved spontaneously or could have been recovered with appropriate treatment within 7 days. Grade 3 infection which could be recovered with appropriate treatment within 7 days. Azacitidine injection site reaction or complications related to azacitidine injection. 2. Febrile neutropenia as defined by CTCAE which could not recovered with appropriate treatment within 7 days. 3. Inability to deliver full dose of volasertib according to the assigned dose level within Cycle 1 due to drug-related AEs. 4. Haematological DLTs. 5. Any other drug-related AEs that resulted in the delay of starting new treatment cycle for ≥4 weeks.
Time Frame: First treatment cycle, up to 28 days
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | Volasertib Monotherapy | Volasertib + Azacitidine Combination
Number analyzed (Participants) | 1 | 0
Participants | 0 |

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Volasertib
Description: The MTD was defined as the highest dose with less than 35% risk of the true dose limiting toxicities (DLT) rate being above 0.33 for schedule A, and the highest dose with less than 40% risk of the true DLT rate being above 0.33 for schedule B. The phase I dose-finding was to be guided by a Bayesian 2-parameter logistic regression model (BLRM) with overdose control in each schedule separately.
Time Frame: First treatment cycle, up to 28 days
Population: Treated Set
Measure: Number; unit: Milligram (mg)/ meter square (m2)
Arm/Group | Volasertib Monotherapy | Volasertib + Azacitidine Combination
Number analyzed (Participants) | 1 | 0
Milligram (mg)/ meter square (m2) | NA — MTD was not determined for this treatment schedule due to premature discontinuation of the trial |

3. Secondary Outcome: Objective Response Defined as Best Overall Response of Complete Remission, Partial Remission or Haematological Improvement According to the International Working Group 2006 Criteria
Description: Objective response defined as best overall response of complete remission, partial remission or haematological improvement according to the International Working Group 2006 criteria. It is based on Complete remission (CR): Bone marrow: <=5% myeloblasts with normal maturation of all cell lines, Peripheral blood: Hemoglobin >=11 Grams Per Decilitre (g/dL), Platelets >=100 x 109/L, Neutrophils >=1.0 x 109/L, Blasts 0%. Peripheral blood responses had to last at least 4 weeks to qualify for CR. Partial remission (PR): All CR criteria if abnormal before treatment except: Bone marrow blasts decreased by >=50% to baseline but still >5%, Cellularity and morphology not relevant. Peripheral blood responses must last at least 4 weeks to qualify for PR. Haematological improvement (HI): HI was evaluated in patients with abnormal pretreatment values based on Erythroid response, Platelet response, Neutrophil response. Peripheral blood responses had to last at least 8 weeks to qualify for HI.
Time Frame: Up to 168 days
Population: Treated Set
Measure: Number; unit: Participants
Arm/Group | Volasertib Monotherapy | Volasertib + Azacitidine Combination
Number analyzed (Participants) | 1 | 0
Participants
  Yes | 0 |
  No | 1 |

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero to the Last Measured Time Point tz of Volasertib (AUC0-tz) (for Monotherapy)
Description: Area under the plasma concentration-time curve over the time interval from zero to the last measured time point tz of volasertib (AUC0-tz) (for monotherapy).
Time Frame: Pharmacokinetic (PK) samples were taken at 5 minutes before drug administration and 0:30, 1:00, 2:00, 3:00, 4:00, 24:00, 167:55, 168:30, 169:00, 169:30, 170:00, 171:00, 172:00, 192:00, 336:00, 504:00, 672:00 hours after drug administration
Population: All evaluable patients were to be included in the PK analysis. Patients who were considered as not evaluable were to be listed with their individual plasma concentrations and individual PK parameters; however, they were not to be included in descriptive statistics for plasma concentrations.
Measure: Number; unit: Nanogram(ng)*hour(h)/milliliter(mL)
Arm/Group | Volasertib Monotherapy
Number analyzed (Participants) | 1
Nanogram(ng)*hour(h)/milliliter(mL)
  Cycle 1 - Day 1 | 2480
  Cycle 1 - Day 8 | 5460

5. Secondary Outcome: Maximum Measured Plasma Concentration of Volasertib (Cmax) (for Monotherapy)
Description: Maximum measured plasma concentration of volasertib (Cmax) (for monotherapy).
Time Frame: PK samples were taken at 5 minutes before drug administration and 0:30, 1:00, 2:00, 3:00, 4:00, 24:00, 167:55, 168:30, 169:00, 169:30, 170:00, 171:00, 172:00, 192:00, 336:00, 504:00, 672:00 hours after drug administration
Population: All evaluable patients were to be included in the Pharmacokinetic (PK) analysis. Patients who were considered as not evaluable were to be listed with their individual plasma concentrations and individual PK parameters; however, they were not to be included in descriptive statistics for plasma concentrations.
Measure: Number; unit: Nanogram(ng)*/milliliter(mL)
Arm/Group | Volasertib Monotherapy
Number analyzed (Participants) | 1
Nanogram(ng)*/milliliter(mL)
  Cycle 1 - Day 1 | 467
  Cycle 1 - Day 8 | 553

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero Extrapolated to Infinity of Volasertib (AUC0-∞) (for Combination)
Description: Area under the plasma concentration-time curve over the time interval from zero extrapolated to infinity of volasertib (AUC0-∞) (for combination).
Time Frame: PK samples were to be taken at 5 minutes before drug administration (167:55) and 168:30, 169:00, 169:30, 170:00, 171:00, 172:00, 192:00, 336:00, 504:00, 672:00 hours after first drug administration of Azacitidine
Population: Due to premature discontinuation of the trial no patient is recruited for combination therapy.
Arm/Group | Volasertib + Azacitidine Combination
Number analyzed (Participants) | 0

7. Secondary Outcome: Maximum Measured Plasma Concentration of Volasertib (Cmax) (for Combination)
Description: Maximum measured plasma concentration of volasertib (Cmax) (for combination).
Time Frame: as for outcome 6
Population: Due to premature discontinuation of the trial no patient is recruited for combination therapy.
Arm/Group | Volasertib + Azacitidine Combination
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after the last dose of study medication, up to 94 days
Arm/Group | Volasertib Monotherapy
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib Monotherapy (N=1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib Monotherapy (N=1)
Cataract (Eye disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Oral lichen planus (Gastrointestinal disorders) | 1
Small intestine ulcer (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Infusion site extravasation (General disorders) | 1
Herpes simplex (Infections and infestations) | 1
Injection site infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Weight decreased (Investigations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Hypertonic bladder (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Trial was prematurely discontinued and only one patient was treated. So it was not possible to draw any conclusion about volasertib monotherapy/with azacitidine, in patients with Myelodysplastic syndrome after Hypomethylating agent treatment failure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.